CLINICAL TRIAL: NCT04787757
Title: Autonomous Robotics for Transcatheter dEliveRy sYstems
Brief Title: Autonomous Robotics for Transcatheter Cardiac Procedures
Acronym: ARTERY
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Politecnico di Milano (Other); Scuola Superiore di Studi Universitari e di Perfezionamento Sant'Anna (Other); KU Leuven (Other); SwissVortex (Unknown); Artiness SRL (Industry); FBGS (Unknown); IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Other Study IDs: ARTERY/08/2021
Record Dates: First submitted 2021-02-26; First posted 2021-03-09 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Mitral Valve Disease; Heart Valve Diseases; Structural Heart Abnormality
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Percutaneous cardiac procedures: Patients undergoing percutaneous cardiac procedures
  Interventions: Procedure: Percutaneous cardiac procedure

INTERVENTIONS:
Procedure: Percutaneous cardiac procedure — Collection and analysis of intraprocedural information to provide artificial intelligence algorithms

SUMMARY:
Cardiovascular diseases represent the most common cause of death worldwide. Percutaneous approaches with intravascular catheters are pivotal, since they allow to treat patients with high perioperative risks. However, catheter-based treatments require steep learning curves and are characterized by poor ergonomics and exposure to damaging radiation. ARTERY will offer a radiation-free approach based on shared-autonomy robotic catheters, with increased user engagement and easy interaction. Intraprocedural three-dimensional echocardiography as well as computed tomography images obtained during usual clinical practice will provide artificial intelligence algorithms that will turn catheter navigation to a simple task. Optical and electromagnetic sensing techniques will ensure a superior view upon the cardiovascular anatomy and will guide the autonomous catheter upon the interventionist supervision, who will be able to take over control at any instant.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* patients admitted to hospital undergoing percutaneous cardiac procedure
* patients able to give informed consent

Exclusion Criteria:

* age <18 years
* refuse to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates to percutaneous cardiac defects repair
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Identification of key procedural elements that will benefit from the technological developments introduced by ARTERY by collecting intraprocedural images | Intraoperative period
  Number of patients undergoing percutaneous cardiac procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita-Salute San Raffaele, Milan, MI, Italy

REFERENCES:
- [Background] Munafo R, Saitta S, Tondi D, Ingallina G, Denti P, Maisano F, Agricola E, Votta E. Automatic 4D mitral valve segmentation from transesophageal echocardiography: a semi-supervised learning approach. Med Biol Eng Comput. 2025 Jan 11. doi: 10.1007/s11517-024-03275-w. Online ahead of print. PMID 39797996